CLINICAL TRIAL: NCT05401695
Title: The Role of Blood Purification by Hemoadsorption as Adjunctive Treatment in Children With Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Tatiya Siripanadorn, MD, Doctor, Chulalongkorn University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ped Critical Care KCMH
Record Dates: First submitted 2022-05-07; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Septic Shock; Multi Organ Failure
Keywords: Blood purification; Hemoperfusion; HA330; PELOD-2 score; PRISM-3 score
MeSH Terms: conditions — Shock, Septic; Multiple Organ Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The historical control group (No Intervention): The historical control group was composed of patients treated septic shock between May 2019 and May 2021. They was received routine treatment for septic shock including intravenous fluid resuscitation, antibiotics, removal of source of infection and inotropic drugs within 6 hours after the diagnosis of sepsis.
- The HA-treated group (Active Comparator): The HA-treated group will be enrolled between July 2021 and May 2022. This group included children with sepsis, who were admitted to our PICU during the study period. All children initially received routine treatment for septic shock as the historical control group. An HA330 disposable hemoperfusion cartridge (HA330; Jafron, Zhuhai City, China) was used with a continuous renal replacement therapy (CRRT) machine (Aquarius® or Primaflex®) in this intervention group.
  Interventions: Device: HA330 hemoadsorption technique

INTERVENTIONS:
Device: HA330 hemoadsorption technique — Hemoadsorption (HA) treatment An HA330 disposable hemoperfusion cartridge (HA330; Jafron, Zhuhai City, China) was used with a continuous renal replacement therapy (CRRT) machine (Aquarius® or Primaflex®) in the intervention group. We will select a blood circuit for each machine according to the patient's body weight. Vascular access will be established with ultrasound-guided insertion of a double-lumen venous catheter into the right internal jugular or femoral vein. HA will be performed for a maximum of 4 hours, and the second session will be started approximately 24 hours after the end of the first session. The blood flow rate will be started low and be gradually increased while monitoring real-time blood pressure and vital signs with an arterial-line monitor. After the end of the HA session, CRRT will be continued if required.
  Arms: The HA-treated group

SUMMARY:
Sepsis is a major healthcare problem and leading cause of death in the pediatric population. Despite advances in supportive care of critically ill patients, sepsis remains an important cause of death worldwide in children. Overall, sepsis incidence peaked in early childhood. There were an estimated 20.3 million incident sepsis cases worldwide among children younger than 5 years. The Surviving Sepsis Campaign (SSC), which standardized the evidence-base approach to management of septic shock and other sepsis-associated organ dysfunction in children, was recently updated. Nevertheless, mortality and costs are still high.

Sepsis is characterized by a complex systemic inflammatory response to a microbial pathogen. A dysregulated host response to infection may result in life-threatening multi-organ dysfunction. Endotoxin, which is found in the outer membrane of Gram-negative bacteria, plays an important role in the pathogenesis of septic shock by producing proinflammatory cytokines. High levels of endotoxin and proinflammatory cytokines are associated with a high mortality rate.

Treatment strategies in sepsis and septic shock include early and adequate fluid resuscitation, vasopressors and inotropic support when indicated, early use of broad-spectrum antibiotics with source control, with close monitoring and organ support, if indicated. Other therapies such as immune-modulation and blood purification have been tried to improve outcomes in patients with sepsis and septic shock. Immunomodulation and blood purification techniques aim at restoring the balance of the immune response to infection, by removing the triggers for the response and the cytokines produced and thereby achieve immune homeostasis. Removing endotoxin and inflammatory cytokines would be an effective adjunctive approach in the management of severe sepsis.

Direct hemoadsorption (HA) is an extracorporeal technique utilized for blood purification. It involves the passage of blood through an adsorption cartridge, where solutes are removed by direct binding to the sorbent material. Over the years, new adsorption cartridge, with improved characteristics have been developed. Resin-directed hemoadsorption is associated with improved oxygenation, hemodynamic status and cardiac function. However, most studies include only adults, and little information is available regarding the clinical experience and efficacy of blood purification for pediatric septic shock.

This pilot study aimed to evaluate the overall clinical outcomes among children who received direct hemoadsorption as an adjunctive treatment for refractory septic shock with high severity scores, compared with outcomes among children admitted to the PICU who received standard treatment.

DETAILED DESCRIPTION:
Study design This pilot study is the prospective interventional cohort study with comparison to a historical control group at a nine-bed PICU at a university referral hospital. Children with septic shock who meet the inclusion criteria will be enrolled. The HA-treated group will be enrolled between July 2021 and May 2022. The historical control group was composed of patients treated between May 2019 and May 2021. Baseline clinical severity scores were matched between the two groups. Investigators will obtained informed consent from the families of all patients. The confounding factor was controlled by matching ratio 1:3 (baseline clinical severity score matching). So sample size of intervention (HA) group was calculate about 10 cases.

Patients The HA group included children with sepsis, as defined by the Surviving Sepsis Campaign guideline 2020, who were admitted to our PICU during the study period. All children initially received routine treatment for septic shock, including intravenous fluid resuscitation, antibiotics, removal of source of infection and inotropic drugs within 6 hours after the diagnosis of sepsis. Patients were included if they: 1) are 30 days to 15 years of age, 2) require any dose of at least one vasopressor and 3) has a Pediatric Logistic Organ Dysfunction (PELOD)-2 score ≥ 10 or Pediatric Risk of Mortality (PRISM)-3 score ≥ 15. Patients receiving end-of-life support, those with uncontrolled bleeding were excluded. The historical control group included patients with sepsis who were admitted to our PICU with the same inclusion criteria and received standard treatment. Patients will be matched according to baseline clinical severity score.

Hemoadsorption (HA) treatment An HA330 disposable hemoperfusion cartridge (HA330; Jafron, Zhuhai City, China) was used with a continuous renal replacement therapy (CRRT) machine (Aquarius® or Primaflex®) in the intervention group. Investigators will select a blood circuit for each machine according to the patient's body weight. For the Aquarius machine, Aqualine S (64-mL blood volume) will be used for body weight < 30 kg and Aqualine (105-mL blood volume) will be used for weight ≥ 30 kg. Four types of blood circuit will be utilized with the Prismaflex machine, including Prismaflex HF20 set (60 mL) for weight < 3-11 kg, Prismaflex M60 set (93 mL) for weight 11-30 kg and Prismaflex M100 set (152 mL) for weight > 30 kg. After rinsing with normal saline solution with heparin, priming the blood circuit and the cartridge with normal saline solution; using 5% albumin or packed red cells (PRC) when the volume of the extracorporeal circuit is more than 10% of the circulatory volume of the patient. If the albumin level is below 3.5 g/dL and hematocrit is above 30%, 5% albumin will be used for priming. If hematocrit is below 30%, PRC will be used. Vascular access will be established with ultrasound-guided insertion of a double-lumen venous catheter into the right internal jugular or femoral vein. The size of the double-lumen catheter is 8 French (Fr) for patients weighing 6-15 kg, 9-10 Fr for those weighing 15-30 kg and 11.5 Fr for those weighing > 30 kg. HA will be performed for a maximum of 4 hours, and the second session will be started approximately 24 hours after the end of the first session. The blood flow rate will be started low and be gradually increased while monitoring real-time blood pressure and vital signs with an arterial-line monitor. After the end of the HA session, CRRT will be continued if required.

Data collection and study endpoints Demographic data, underlying disease and source of infection are extracted from patients' hospital charts. Blood gas data, type of respiratory support, dose of vasopressors and laboratory data will be recorded at baseline, 24 hours, 48 hours and 72 hours. The baseline is define as a time before HA treatment in the intervention group and when patients will be noted to have no response to initial resuscitation in the control group. The severity of organ dysfunction or failure will be expressed with the PELOD-2 score and PRISM-3 score and recorded at the four time points above. The dose of vasoactive/vasopressor agents will be expressed as the vasoactive inotropic score (VIS), calculated as: dopamine dose + dobutamine dose + (epinephrine dose × 100) + (norepinephrine dose × 100) + (milrinone dose × 10) + (vasopressin dose × 10,000), with doses expressed as mcg/kg/min for most drugs and as U/kg/min for vasopressin. The primary endpoints are the reduction in PELOD-2 and PRISM-3 scores at 72 hours, with adjustment for baseline between the HA and control groups. The secondary endpoints are the reductions in IL-6, VIS, oxygenation index, serum creatinine, base excess and lactate at 72 hours; length of PICU stay, hospital stay and mechanical ventilation; and 28-day mortality.

Laboratory methods Serum samples are analyzed by Direct Ion Selective Electrode for arterial blood gas analysis, which include the data of arterial lactate, base excess and oxygenation index. Complete blood count (CBC) are analyzed by Chemical dye, Laser scattering, SF Cube, Sheath Fluid and Impedance Method to evaluated white blood cell count (WBC) and platelets. Serum creatinine (Cr) and other blood chemistry are analyzed by Reflotron method. IL-6 is analyzed by Electrochemiluminescence immunoassay (ECLIA).

Data analysis and statistics Data analysis using the median with range (minimum-maximum) or mean ± standard deviation. Investigators will use Student's t-test analysis for continuous variables data and Fisher's exact test for categorical variables data. Within-group analysis of PELOD-2, PRISM-3, oxygenation index, VIS, creatinine, base excess, endotoxin levels and lactate will be performed with paired t-tests; between-group comparisons are performed with analysis of covariance (ANCOVA) at 72 hours, with adjustment for the baseline in each group.

ELIGIBILITY:
Inclusion Criteria:

Children were 30 days to 15 years of age, who required any dose of at least one vasopressor and one of following

1. Pediatric Logistic Organ Dysfunction (PELOD)-2 score ≥ 10
2. Pediatric Risk of Mortality (PRISM)-3 score ≥ 15

Exclusion Criteria:

1. Patients receiving end-of-life support
2. Patients who uncontrolled bleeding

Ages: 1 Month to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
The reduction of PELOD-2 score | At 72 hours after start treatment
  The PELOD-2 score, Pediatrics Logistic Organ Dysfunction-2 score as a descriptive scoring system for organ dysfunction. It consists of 10 variables which represent 5 organ dysfunctions. A higher PELOD-2 score correlates with a higher number of organ failures and mortality rate. The minimum of PELOD-2 score is zero, which mortality rate is 0.4%. The higher PELOD-2 score more than 16.8 correlated with mortality rate >60%.
The reduction of PRISM-3 score | At 72 hours after start treatment
  The PRISM-3 score, Pediatrics Risk of Mortality-3 score has 17 physiologic variables subdivided into 26 ranges. Similar to the PELOD-2 score, the higher PRISM-3 score correlates with a higher number of organ failures and mortality rate. The minimum of PRISM-3 score is zero. The maximum PELOD-2 score is 76.

SECONDARY OUTCOMES:
The reduction in IL-6 | At 72 hours after start treatment
The reduction in VIS at 72 hours | At 72 hours after start treatment
  Vasoactive inotropic score (VIS)
The reduction in lactate levels at 72 hours | At 72 hours after start treatment
The reduction in oxygenation index at 72 hours | At 72 hours after start treatment
The length of PICU stay | Assessed up to 2 years after PICU admission
The length of hospital stay | Assessed up to 2 years after admission in hospital
The length of mechanical ventilation | Assessed up to 2 years after the first intubation in PICU
The 28-day mortality | 28 days from admission

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No